CLINICAL TRIAL: NCT00764647
Title: Evaluation of Education Program for Family Caregivers of Frail Elders
Brief Title: Education Program for Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Barbara Nunley, PhD, Associate Professor Faculty Emerita, West Virginia University School of Nursing., CAMC Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-02-1779
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Stress
Keywords: family caregivers; caregiver education; caregiver burden; caregiver hardiness; caregiver depressive symptoms
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Education program for family caregivers of frail elders.
  Interventions: Behavioral: Education program for family caregivers of frail elders

INTERVENTIONS:
Behavioral: Education program for family caregivers of frail elders — Family caregiver participants in the educational program will receive an educational course presented by the investigator that focuses on the care of the frail elder and themselves. The course will involve four to five consecutive weekly sessions, each 2 1/2 to 3 hours long. The educational program will be offered biannually, spring and fall seasons.

SUMMARY:
The purpose of this evaluation was to determine the effectiveness of an educational program designed to assist family caregivers to learn the knowledge and skills to take better care of their frail elder relatives and themselves.

DETAILED DESCRIPTION:
Spouses, children, and other family members typically care for frail elderly persons. These family caregivers attempt to provide care for their relative in the home, despite the potential for excessive stress to themselves. This care may extend over many years, involving unrelenting management of their relative, which puts the caregiver at risk for the development of physical and mental health consequences. The stress of caring for a frail elder may result in the institutionalization of the care receiver due to declining health or abilities in the caregiver as caregivers frequently continue to provide care at the expense of their own health. The goal of the education program is to fill an important need, that is, assist caregivers to become empowered, hardier, and have the ability to cope with the stress associated with caregiving. The aim is to investigate whether this educational intervention improves selected outcomes for family caregivers of frail elders. The selected outcomes are knowledge of caregiving, hardiness, quality of life, physical health, depressive symptoms, burden, and coping.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* family member participating in care of a frail elder (60 years and older)

Exclusion Criteria:

* unable to speak or read English (materials are written in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Hardiness (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  Hardiness was measured using the Psychological Hardiness Scale, a 40 item scale (Younkin & Betz, 1996). Responses for each item were obtained on a 5-point Likert continuum from "Strongly Disagree" (1) to Strongly Agree (5).

SECONDARY OUTCOMES:
Knowledge of Caregiving (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  Knowledge about caregiving was operationalized by total score on a content-specific test (17 items) for the family caregivers' educational program that measured knowledge and behaviors. True/false answers were given to items.
Quality of Life (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  Quality of life measured using a Cantril (1965) ladder scale. The participants viewed a picture of a ladder with nine rungs, with the top rung labeled "best possible life" (9) and the bottom rung labeled "worst possible life (0).
Physical and Mental Health (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  The SF-36v2 Health Survey (Ware & Sherboume, 1992), a 36-item self-report scale was used to measure the caregiver's view of their health.
Depressive Symptomatology (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  The Center for Epidemiologic Studies-Depression Scale (CES-D; Radloff, 1977), a 20 item self report scale, was used to measure depressive symptomatology. Participants rated how frequently each symptom occurred during the past week on a scale ranging from rarely or none of the time (0) to most or all of the time (3).
Caregiver Burden (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  The Caregiver Burden Inventory (CBI), developed by Novak and Guest (1989), a 24-item multidimensional measure was used to measure caregiver burden. This inventory includes five factors: Time-dependence burden, Developmental burden, physical burden, Social burden, and Emotional burden.
Coping (change over time) | pre-intervention, immediate post-intervention, six-month post-intervention, and twelve-month post intervention
  The Jalowiec Coping Scale (JCS) (Jalowiec, Murphy, & Powers, 1984) was used to measure coping mechanisms. There are 60 items classified into 8 different coping styles: confrontive, evasive, optimistic, fatalistic, emotive, palliative, supportant, and self-reliant.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Nunley, PhD, RN, Principal Investigator — West Virginia University School of Nursing
Locations (1):
- West Virginia University Robert C. Byrd Health Sciences Center, Charleston Division, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorensen S, Pinquart M, Duberstein P. How effective are interventions with caregivers? An updated meta-analysis. Gerontologist. 2002 Jun;42(3):356-72. doi: 10.1093/geront/42.3.356. PMID 12040138
- [Background] Burgio L, Lichstein KL, Nichols L, Czaja S, Gallagher-Thompson D, Bourgeois M, Stevens A, Ory M, Schulz R; REACH Investigators. Judging outcomes in psychosocial interventions for dementia caregivers: the problem of treatment implementation. Gerontologist. 2001 Aug;41(4):481-9. doi: 10.1093/geront/41.4.481. PMID 11490046
- [Background] Acton GJ, Kang J. Interventions to reduce the burden of caregiving for an adult with dementia: a meta-analysis. Res Nurs Health. 2001 Oct;24(5):349-60. doi: 10.1002/nur.1036. PMID 11746065